CLINICAL TRIAL: NCT05366400
Title: Evaluation of the Relationship Between Right Atrial Volume Index, Functional Capacity and Inflammatory Biomarkers in Patients With Chronic Obstructive Lung Disease and Right Heart Affection.
Brief Title: Relationship Between Right Atrial Volume Index, Functional Capacity and Inflammatory Biomarkers in Patients With COPD.
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Other Study IDs: RAVI in COPD patients
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: COPD; Right Heart Failure
Keywords: Chronic obstructive lung disease.; Right atrial volume index.; Functional capacity.; Adiponectin.; Hs-CRP.; IL1b.; Neoptrin.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (CAT) ≥ 10: CAT is an eight-item questionnaire with a six-item Likert scale ranging from 0 to 5. The score ranges from zero (completely asymptomatic) to 40 (extremely symptomatic). A CAT score ≥10 is associated with a significantly impaired health status.
  Interventions: Diagnostic Test: ECHO
- Group II (CAT) < 10: CAT is an eight-item questionnaire with a six-item Likert scale ranging from 0 to 5. The score ranges from zero (completely asymptomatic) to 40 (extremely symptomatic). A CAT score < 10 is associated with a significantly preserved health status.
  Interventions: Diagnostic Test: ECHO

INTERVENTIONS:
Diagnostic Test: ECHO — Conventional routine tests and ECHO will be assessed. Biomarkers will be measured using ELISA The functional capacity was assessed by the COPD assessment test (CAT) questionnaire.

SUMMARY:
Right ventricular (RV) dysfunction is associated with increased morbidity and mortality in patients with chronic obstructive pulmonary disease (COPD). Assessment of RV function by echocardiography is challenging. Easy visualization of the right atrium (RA) by echocardiography , allows quantitative, highly reproducible assessment of RA volume. The aim of the present study is to evaluate the relationship between the right atrial volume index (RAVI) and functional capacity in patients with COPD , quantified by the COPD assessment test (CAT) questionnaire as an early predictor of right heart affection.

DETAILED DESCRIPTION:
1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. All participants agreed to take part in this clinical study and provide informed consent.
3. Patients who were selected from patients visited Chest Department or attending Chest outpatient clinic of Tanta University Hospitals, Echocardiography was done in the Cardiology Department..
4. Complete physical and laboratory assessment will be done for all patients.
5. Serum samples will be collected for measuring the biomarkers.
6. 150 patients with COPD and preserved left ventricular systolic function, ejection fraction (LVEF) > 55% will enrolled. The RA volume calculated by biplane area length method using four chamber view twice and indexed to body surface area (RAVI). Assessment of RV systolic function was done using tricuspid annular plane systolic excursion (TAPSE), and peak systolic velocity (S'tri) using tissue Doppler imaging at the tricuspid annulus. The functional capacity was assessed by the COPD assessment test (CAT) questionnaire.
7. For each participant, blood samples were obtained and levels of adiponectin, IL-1B, high-sensitivity C-reactive protein and Neopterin will be determined in all studied subjects.
8. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion criteria - Patients included were > 18 years old of both sexes and left ventricular ejection fraction (LVEF) >55%.The following clinical and demographic parameters were recorded; age, sex, Current cigarette smoking was defined as active smoking within the past 12 months. Coronary artery disease was obtained by history or previous medical records.

Exclusion criteria

- Patients with diagnosis of other respiratory diseases (e.g. asthma, interstitial pulmonary fibrosis , tuberculosis or lung cancer ), ischemic heart disease, congestive heart failure, valvular heart disease and congenital heart diseases, were excluded. Other chronic diseases, such as kidney or liver failure and cancer were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All COPD patients participate in this study, were diagnosed on clinical based data and confirmed by spirometry findings according to the diagnostic criteria of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines.
  This study was carried out on COPD patients who were selected from patients visited Chest Department or attending Chest outpatient clinic of Tanta University Hospitals, Echocardiography was done in the Cardiology Department.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
RAVI (ml/m2) | 3 month
  Right atrial volume index
Adiponectin (mg/L) | 3 month
  Serum Level
Neopterin (nmol/L) | 3 month
  Serum Level
IL-1beta (pg/mL) | 3 month
  Serum Level

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Principal Investigator — Damanhour University; Lamiaa Khedr, Ass. Prof., Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thierer J, Acosta A, Vainstein N, Sultan M, Francesia A, Marino J, Prado AH, Guglielmone R, Trivi M, Boero L, Brites F, Anker S. Relation of left ventricular ejection fraction and functional capacity with metabolism and inflammation in chronic heart failure with reduced ejection fraction (from the MIMICA Study). Am J Cardiol. 2010 Apr 1;105(7):977-83. doi: 10.1016/j.amjcard.2009.11.017. Epub 2010 Feb 13. PMID 20346316
- [Background] de Groote P, Millaire A, Foucher-Hossein C, Nugue O, Marchandise X, Ducloux G, Lablanche JM. Right ventricular ejection fraction is an independent predictor of survival in patients with moderate heart failure. J Am Coll Cardiol. 1998 Oct;32(4):948-54. doi: 10.1016/s0735-1097(98)00337-4. PMID 9768716